CLINICAL TRIAL: NCT03253523
Title: Post-traumatic Occipital Neuralgia - Surgical Versus Medical Management
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients did not want to take part in the experimental arm of the study as all have opted for the current standard of care procedure.
Sponsor: Rush University Medical Center (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00148116
Record Dates: First submitted 2017-08-15; First posted 2017-08-18 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Post-Traumatic Neuralgia; Occipital Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continued maximal medical management (No Intervention)
- Surgical occipital nerve neurolysis (Experimental)
  Interventions: Procedure: Occipital neurolysis

INTERVENTIONS:
Procedure: Occipital neurolysis — Surgical occipital nerve decompression
  Arms: Surgical occipital nerve neurolysis

SUMMARY:
Occipital neuralgia and subsequent headaches are associated with significant morbidity and impact quality of life and ability to work. Treatment is primarily medical and consists of non-steroidal anti-inflammatory medications and medications to treat neuropathic pain. Many patient exhaust medical management options and suffer from persistent symptoms.

Surgical management of chronic headaches including occipital neuralgia is emerging as a tool to relieve pain and the burden of morbidity associated with this condition. Dr. Bahman Guyuron has been reporting positive results in the literature for the past 20 years. In a systematic review of 14 papers it has been demonstrated that peripheral nerve surgery for migraines is effective and leads to an improvement of symptoms for 86% of patients. Complication rates were low across all studies included. Additionally, Dr Ivica Ducic has reported success specifically treating occipital neuralgia headaches, with significant improvements in subjective pain outcomes post-operatively. The mechanism behind this is thought to be similar to carpal tunnel syndrome, whereby peripheral nerve compression causes nerve irritation and pain. The ensuing inflammatory response to tissue injury can cause sensitization of nociceptors, resulting in hyperalgesia or allodynia. Surgical release of tight surrounding soft tissues results in nerve decompression and relief of symptoms.

Although there are multiple case series and empiric evidence supporting the safety and efficacy of occipital migraine surgery, there are no randomized controlled studies comparing surgical intervention with continued medical management.

As part of the present study, the investigators intend to randomize patients who have exhausted maximal medical treatment of post-traumatic occipital headaches to either a surgical management group or a continued medical management group. Surgical intervention will consist of neurolysis, or release, of the occipital nerves.

ELIGIBILITY:
Inclusion Criteria:

* History of head or neck trauma as an inciting event for occipital headaches
* Occipital neuralgia headache, as diagnosed by neurologist, and as defined by the International Classification of Headache Disorders (ICHD-3). 13.4 - occipital neuralgia:

Description:

Unilateral or bilateral paroxysmal, shooting or stabbing pain in the posterior part of the scalp, in the distribution of the greater, lesser or third occipital nerves, sometimes accompanied by diminished sensation or dysaesthesia in the affected area and commonly associated with tenderness over the involved nerve(s).

Diagnostic criteria:

* Unilateral or bilateral pain fulfilling criteria B-E
* Pain is located in the distribution of the greater, lesser and/or third occipital nerves
* Pain has two of the following three characteristics:

  * recurring in paroxysmal attacks lasting from a few seconds to minutes
  * severe intensity
  * shooting, stabbing or sharp in quality
* Pain is associated with both of the following:

  * dysaesthesia and/or allodynia apparent during innocuous stimulation of the scalp and/or hair
* either or both of the following:

  * tenderness over the affected nerve branches
  * trigger points at the emergence of the greater occipital nerve or in the area of distribution of C2
* Pain is eased temporarily by local anaesthetic block of the affected nerve
* Not better accounted for by another ICHD-3 diagnosis.

Comments:

The pain of 13.4 Occipital neuralgia may reach the fronto-orbital area through trigeminocervical interneuronal connections in the trigeminal spinal nuclei.

13.4 Occipital neuralgia must be distinguished from occipital referral of pain arising from the atlantoaxial or upper zygapophyseal joints or from tender trigger points in neck muscles or their insertions.

* Age: 18-65
* Male and female

Exclusion Criteria:

* Headache of any etiology other than specified in the inclusion criteria.
* Patients with occipital referral of pain arising from the atlantoaxial or upper zygapophyseal joints or from tender trigger points in neck muscles or their insertions
* Pregnant or breastfeeding females
* Patients with significant comorbidities including short life expectancy, malignancy, degenerative central nervous system diseases, infection, severe psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Average visual analogue scale of pain intensity | 6 months
  Assess patient's average headache on a visual analog scale from 1-10, 10 being the worst pain
Headache days per month | 6 months
  Assess patient-reported number of days with headaches per month, in days
Duration of average headache | 6 months
  Assess patient-reported average duration of headaches, in hours
Change in Migraine Headache Index (the multiple of scores 1-3) at 6 months | from baseline to 6 months
  The Migraine Headache Index (MHI) is a commonly used metric in the plastic and reconstructive surgery literature to assess pre- and postoperative headache severity. The score is a product of headache duration (in days), frequency (in days per month), and severity (on a scale from 1 to 10). The score ranges from 0 to 300, with higher scores corresponding to worse migraine symptoms. Change in MHI score between pre-operative and 6-month postoperatively will be assessed.

SECONDARY OUTCOMES:
Subjective patient recorded outcomes of quality of life | 6 months
  Assessment of quality of life using the Headache Impact Test (HIT-6) tool. The scores range from 36 to 78, with scores over 50 indicating some degree of impact of headaches on quality of life.
Medication intake | 6 months
  Patient-reported average intake of analgesic medications for occipital neuralgia pain
Engagement in activity pre- and post-operatively | 6 months
  Patient-reported ability to return to daily work and recreational activities. Outcome will be measured in days per month when patient stays home and is unable to work or otherwise engage in recreational activities secondary to migraine symptoms.
Patient satisfaction | 6 months
  Reported as the number of patients that answer "Yes" to question: 'Would you have the surgery again?'

CONTACTS AND LOCATIONS:
Overall Officials: Amir Dorafshar, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States